CLINICAL TRIAL: NCT03069014
Title: A 6-months Prospective, Multi-center, Double-blind, Placebo-controlled, Randomized, Adaptive-trial-design Study to Evaluate Safety, Tolerability and Exploratory Endpoints of Either Placebo or Two Different Oral Doses of LM11A-31-BHS in Patients With Mild to Moderate Probable Alzheimer's Disease
Brief Title: Study of LM11A-31-BHS in Mild-moderate AD Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PharmatrophiX Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSC15001; 2015-005263-16 (EudraCT Number); 1R01AG051596-01A1 (NIH)
Record Dates: First submitted 2017-02-03; First posted 2017-03-03 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Mild to Moderate Alzheimer's Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 400mg LM11A-31-BHS (Active Comparator): 400mg LM11A-31-BHS and 400mg Placebo per day
  Interventions: Drug: 400mg LM11A-31-BHS; Drug: Placebos
- 800mg LM11A-31-BHS (Active Comparator): 800mg LM11A-31-BHS
  Interventions: Drug: 800mg LM11A-31-BHS
- Placebos (Placebo Comparator): 800mg (microcrystalline cellulose with 0.5 - 1% magnesium stearate) per day
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: 400mg LM11A-31-BHS — 1 Oral Capsules (200mg of LM11A-31-BHS and 200mg of placebo) twice daily (morning & evening) for 26 weeks
  Arms: 400mg LM11A-31-BHS
Drug: 800mg LM11A-31-BHS — 2 Oral Capsules (200mg of LM11A-31-BHS) twice daily (morning & evening) for 26 weeks
  Arms: 800mg LM11A-31-BHS
Drug: Placebos — 2 Oral Capsules (200mg of Placebo) twice daily (morning & evening) for 26 weeks
  Arms: 400mg LM11A-31-BHS; Placebos

SUMMARY:
The purpose of this study is to determine the safety of 2 doses of LM11A-31-BHS in 180 patients with Alzheimer's Disease versus placebo and to access biomarker and clinical exploratory endpoints of LM11A-31-BHS

DETAILED DESCRIPTION:
The goal of this AD Pilot is to conduct a prospective, double-blind, multicenter, phase IIa exploratory safety, feasibility and proof-of-concept trial in mild to moderate Alzheimer's disease patients with the orally bioavailable p75 neurotrophin receptor ligand LM11A-31-BHS dosed twice daily for 26 weeks. Successful completion of this trial will provide the safety, endpoint and statistical basis for the design and execution of a phase 2b/3 efficacy trial. It will also bring to the AD field a much-needed new set of target mechanisms and will help pioneer the strategy of the concomitant targeting of multiple fundamental AD-related pathological processes.

During the 26 weeks study period the eligible patients will be invited to 5 visits.

Safety monitoring will include the full extent of phase 2 clinical, electrophysiological and laboratory testing.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (non-childbearing potential) with a diagnosis of Alzheimer's disease according to McKhann (2011) criteria
2. Age 50-85 years (50-80 in Czech Republic)
3. MRI or CT assessment within six months before baseline, corroborating the clinical diagnosis of AD and excluding other potential causes of dementia, especially cerebrovascular lesions (see exclusion criteria, number 3)
4. CSF AD specific biomarker profile; positive, defined as CSF Aβ42 < 550 ng l-1 or an Aβ 40/42 ratio < 0.89
5. Mild to moderate stage of Alzheimer's disease according to MMSE ≥ 18 and ≤ 26
6. Absence of major depressive disease according to GDS of < 5
7. Modified Hachinski Ischemic Scale ≤ 4
8. Formal education for eight or more years
9. Previous decline in cognition for more than six months as documented in patient medical records
10. A caregiver available and living in the same household or interacting with the patient a sufficient time each week (in Czech Republic: providing personal care for the patient during at least 10 hours per week ) and available if necessary to assure administration of drug
11. Patients living at home or nursing home setting without continuous nursing care
12. General health status acceptable for a participation in a 6-month clinical trial
13. Ability to swallow capsules
14. Stable pharmacological treatment of any other chronic condition for at least one month prior to screening
15. Stable treatment with one of the acetylcholinesterase inhibitors donepezil (Aricept ®), galantamine (Razadyne®), or rivastigmine (Exelon) or the partial NMDA receptor antagonist with memantine (Namenda®) at least 3-months before baseline Visit or Combination of both treatments mentioned above
16. No regular intake of prohibited medications as noted in Section 11.8 of the protocol
17. Signed informed consent by the patient, examined and verified to be mentally capable by an independent physician, prior to the initiation of any study specific procedure. Signed consent of the caregiver (see inclusion criteria 10).

Exclusion Criteria:

1. Failure to perform screening or baseline examinations
2. Hospitalization or change of chronic concomitant medication one month prior to screening or during screening period
3. Clinical, laboratory or neuro-imaging findings consistent with:

   * Other primary degenerative dementia, (dementia with Lewy bodies, fronto-temporal dementia, Huntington's disease, Creutzfeldt-Jakob Disease, Down's syndrome, etc.)
   * Other neurodegenerative condition (Parkinson's disease, amyotrophic lateral sclerosis, etc.)
   * Cerebrovascular disease (major infarct, one strategic or multiple lacunar infarcts, extensive white matter lesions > one quarter of the total white matter)
   * Other central nervous system diseases (severe head trauma, tumors, subdural hematoma or other space occupying processes, etc.)
   * Seizure disorder
   * Other infectious, metabolic or systemic diseases affecting central nervous system (syphilis, present hypothyroidism, present vitamin B12 or folate deficiency, serum electrolytes out of normal range, juvenile onset diabetes mellitus, etc.)
4. A current DSM-IV diagnosis of active major depression, schizophrenia or bipolar disorder
5. Clinically significant, advanced or unstable disease that may interfere with primary or secondary variable evaluations, and which may bias the assessment of the clinical or mental status of the patient or put the patient at special risk, such as:

   * chronic liver disease, liver function test abnormalities or other signs of hepatic insufficiency (ALT, AST, Gamma GT, alkaline phosphatase > 2.5 ULN)
   * Respiratory insufficiency
   * Renal insufficiency (serum creatinine > 2mg/dl) or creatinine clearance ≤ 30 mL/min according to Cockcroft-Gault formula). In case of creatinine clearance ≤ 30mL/min, an alternative verification of the renal function must be completed using Cystatin C analysis. In case of normal level of Cystatin C, the patient can be included
   * Heart disease (myocardial infarction, unstable angina, heart failure, Cardiomyopathy within six months before screening)
   * Bradycardia (heart beat < 50/min.) or tachycardia (heart beat > 95/min.)
   * Hypertension (> 180/95 / Czech Republic >160/95) or hypotension (< 90/60) requiring treatment with more than three drugs
   * AV block (type II / Mobitz II and type III), congenital long QT syndrome, sinus node dysfunction or prolonged QTcB-interval (males > 450 and females > 470 msec.)
   * Uncontrolled diabetes defined by HbA1c > 8.5
   * Malignancies within the last five years except skin malignancies (other than melanoma) or indolent prostate cancer
   * Metastases
6. Disability that may prevent the patient from completing all study requirements (e.g. blindness, deafness, severe language difficulty, etc.)
7. Women who are fertile and of childbearing potential
8. Chronic daily drug intake of ≥ 14 days or expected for ≥ 14 days:

   * benzodiazepines (except lorazepam ≤ 1mg for sleeping disorders only), neuroleptics or major sedatives
   * Antiepileptics
   * Centrally active anti-hypertensive drugs (clonidine, l-methyl DOPA, guanidine, guanfacine, etc.)
   * Opioid containing analgesics
9. Nootropic drugs with exception of Ginko Biloba
10. Suspected or known drug or alcohol abuse, i.e. more than approximately 60 g alcohol (approximately 1 liter of beer or 0.5 liter of wine / in Czech Republic: 20 g alcohol per day for females (500 ml of beer or 250 ml of wine) and 30g alcohol per day for males (approximately 750 ml of beer or 375 ml of wine)) per day indicated by elevated MCV significantly above normal value at screening
11. Suspected or known allergy to any components of the study treatments
12. Enrollment in another investigational study or intake of investigational drug within the previous three months
13. Any condition, which, in the opinion of the investigator, makes the patient unsuitable for inclusion
14. If patient is in any way dependent on the sponsor or the principal investigator or if the patient is accommodated in an establishment on judicial or administrative order

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Number of AEs/SAEs within the 26-week study period | 26 weeks
  number of subjects with AEs/SAEs, changes in vital signs and laboratory examinations

SECONDARY OUTCOMES:
Statistically relevant changes in CSF-Biomarkers between baseline and final visit | 26 weeks
  CSF-Biomarkers (tau, ptau, Aβ40, Aβ42, AchE activity)
Statistically relevant changes in working memory ability between baseline and final visit assessed with the Controlled Oral Word Association Test (COWAT) | 26 weeks
  Controlled Oral Word Association Test (COWAT)
Statistically relevant changes in word fluency between baseline and final visit assessed with the Category Fluency Test (CFT) | 26 weeks
  Category Fluency Test (CFT)
Statistically relevant changes in processing speed between baseline and final visit assessed with the Coding Test (Subtest of the Wechsler Adult Intelligence Scale) | 26 weeks
  Coding Test (Subtest of the Wechsler Adult Intelligence Scale)
Statistically relevant changes in executive functions between baseline and final visit assessed with the Digit Span test (Subtest of the Wechsler Adult Intelligence Scale) | 26 weeks
  Digit Span test (Subtest of the Wechsler Adult Intelligence Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Windisch, PhD, Principal Investigator — NeuroScios GmbH
Locations (21):
- Austria (2):
  - University Hospital Graz, Graz, Styria
  - Landeskrankenhaus Hall, Hall in Tirol, Tyrol
- Czechia (4):
  - Vestra clinics s.r.o, Rychnov nad Kněžnou, Kralovehadrecky Kraj
  - NEUROHK s.r.o, Choceň, Pardubický kraj
  - Charles University, Prague, Prague
  - Neurology Clinic of Martin Urbanek, Brno, South Moravian
- Germany (9):
  - Nordwestkrankenhaus Sanderbusch, Sande, Friesland
  - Zentrum für klinische Forschung, Bad Homburg, Hesse
  - Studienzentrum Nordwest, Westerstede, Lower Saxony
  - Universitätsklinik Magdeburg, Klinik für Neurologie, Magdeburg, Sachsen Anthal
  - Sächsisches Krankenhaus Arnsdorf, Arnsdorf, Saxony
  - Pharmakologisches Studienzentrum Chemnitz GmbH, Chemnitz, Saxony
  - Charité Universitätsmedizin Berlin, Berlin
  - Neurologie Sendlinger Strasse Studien- und Gedächtniszentrum München, München
  - LMU München Klinik für Psychiatrie und Psychotherapie, München
- Spain (5):
  - Fundació ACE, Barcelona, Catalonia
  - Fundación de Gestión Sanitaria del Hospital de la Santa Creu I Sant Pau, C, Barcelona, Catalonia
  - Hospital Clínic de Barcelona, Barcelona, Catalonia
  - Hospital la Paz, Madrid
  - Hospital Virgen del Rocío, Seville
- Karolinska University, Stockholm, Stockholms Iän, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shanks HRC, Chen K, Reiman EM, Blennow K, Cummings JL, Massa SM, Longo FM, Borjesson-Hanson A, Windisch M, Schmitz TW. p75 neurotrophin receptor modulation in mild to moderate Alzheimer disease: a randomized, placebo-controlled phase 2a trial. Nat Med. 2024 Jun;30(6):1761-1770. doi: 10.1038/s41591-024-02977-w. Epub 2024 May 17. PMID 38760589
- [Derived] Liu G, He M, Wu C, Lv P, Sun H, Wang H, Xin X, Liao H. Axonal injury mediated by neuronal p75NTR/TRAF6/JNK pathway contributes to cognitive impairment after repetitive mTBI. Exp Neurol. 2024 Feb;372:114618. doi: 10.1016/j.expneurol.2023.114618. Epub 2023 Nov 27. PMID 38029807
- [Derived] Malik SC, Sozmen EG, Baeza-Raja B, Le Moan N, Akassoglou K, Schachtrup C. In vivo functions of p75NTR: challenges and opportunities for an emerging therapeutic target. Trends Pharmacol Sci. 2021 Sep;42(9):772-788. doi: 10.1016/j.tips.2021.06.006. Epub 2021 Jul 29. PMID 34334250